CLINICAL TRIAL: NCT03215680
Title: Assessment of Impact of High Temperature Climate on Urinary Iodine Concentration in Women of Reproductive Age
Brief Title: Climat Impact on Urinary Iodine Concentration
Acronym: LION
Status: Completed | Type: Observational
Sponsor: Swiss Federal Institute of Technology (Other)
Collaborators: Ministry of Health, Tanzania (Other Government); North-West University, South Africa (Other)
Responsible Party: Principal Investigator, Prof. Michael B. Zimmermann, Prof. Dr., Swiss Federal Institute of Technology
Other Study IDs: LION
Record Dates: First submitted 2017-07-10; First posted 2017-07-12 (Actual); Last update posted 2021-03-26 (Actual); Status verified 2021-03

CONDITIONS: Iodine Deficiency
Keywords: Urinary iodine concentration
MeSH Terms: interventions — Climate

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — 24h urine samples, spot urine samples, dried blood spots
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Tanzanian Women of Reproductive Age: Healthy women of reproductive age living in Tanzania in an area with hot and temperate climate
  Interventions: Other: Climate
- South African Women of Reproductive Age: Healthy women of reproductive age living in South Africa in an area with hot and temperate climate
  Interventions: Other: Climate

INTERVENTIONS:
Other: Climate — Hot and temperate climate

SUMMARY:
Urinary iodine concentration (UIC) is the recommended biomarker of iodine status in populations. Yet, the influence of climate on UIC remains unclear. Hot climate may reduce urine volume and consequently increase UIC independent of iodine status. This could lead to an overestimation of population iodine intake, thus masking iodine deficiency in vulnerable groups.

In this longitudinal observational cohort study in women of reproductive age we will collect 24h and spot urine samples in the summer and winter season. The influence of high temperature climates on UIC, measured and estimated urinary iodine excretion will be estimated.

ELIGIBILITY:
* Female
* Non-pregnant and non-lactating
* General good health, assessed by no reported treatment for chronic disease
* Non-smoking
* No known history of major medical illnesses or thyroid dysfunction as well as gastrointestinal or metabolic disorders and taking no chronic medication
* Residence at the respective study site for 12 months or longer and no plans of moving away during the study year.
* No use of iodine containing dietary supplements during the last 6 months
* No use of X-ray / CT contrast agent or iodine containing medication within the last year
* No use of iodine containing disinfectants during the last 6 months
* Participants should be between 18 and 49 years at date of enrollment

Ages: 18 Years to 49 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Healthy women between 18 and 49 years of age
Sampling Method: Non-Probability Sample
Enrollment: 363 (Actual)
Dates: Start 2017-07-10 (Actual); Primary Completion 2018-12-31 (Actual); Study Completion 2018-12-31 (Actual)

PRIMARY OUTCOMES:
Urinary iodine concentration | 6 months
  Measured in 24h urine collections

SECONDARY OUTCOMES:
Urinary iodine excretion | 6 months
  Measured in 24 h urine collections

OTHER OUTCOMES:
Urinary iodine concentration | 6 months
  Measured in spot urine samples
Urinary iodine excretion | 6 months
  Measured in spot urine samples

CONTACTS AND LOCATIONS:
Overall Officials: Michael B Zimmermann, Prof. Dr., Principal Investigator — ETH Zurich
Locations (2):
- Centre of Excellence for Nutrition, Faculty of Health Science, North West University, Potchefstroom, South Africa
- Ministry of Health, Community Development Gender, Elderly and Children, Dar es Salaam, Tanzania

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Arns-Glaser L, Zandberg L, Assey VD, Baumgartner J, Abdallah F, Galetti V, Dary O, Zimmermann MB, Andersson M. Seasonal effects on urinary iodine concentrations in women of reproductive age: An observational study in Tanzania and South Africa. Am J Clin Nutr. 2022 Jan 11;115(1):298-309. doi: 10.1093/ajcn/nqab327. PMID 34601579